CLINICAL TRIAL: NCT07046559
Title: A Single- and Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY4066708 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 27332; J5Z-MC-OTAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-05-13; First posted 2025-07-01 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (15):
- Part A Cohort 1: Single-Ascending Dose (SAD)- LY4066708 (Experimental): LY4066708 administered by intravenous (IV) injection
  Interventions: Drug: LY4066708
- Part A Cohort 2: SAD- LY4066708 (Experimental): LY4066708 administered by IV injection
  Interventions: Drug: LY4066708
- Part A Cohort 3A: SAD- LY4066708 (Experimental): LY4066708 administered by subcutaneous (SC) injection
  Interventions: Drug: LY4066708
- Part A Cohort 3B: SAD- LY4066708 (Experimental): LY4066708 administered by SC injection
  Interventions: Drug: LY4066708
- Part A Cohort 4: SAD- LY4066708 (Experimental): LY4066708 administered by IV injection
  Interventions: Drug: LY4066708
- Part A Cohort 5: SAD- LY4066708 (Experimental): LY4066708 administered by IV injection
  Interventions: Drug: LY4066708
- Part A Cohort 5A: SAD- LY4066708 (Experimental): LY4066708 administered by IV injection
  Interventions: Drug: LY4066708
- Part A Cohort 6A: SAD- LY4066708 (Experimental): LY4066708 administered by IV injection
  Interventions: Drug: LY4066708
- Part A Cohort 6: SAD- LY4066708 (Experimental): LY4066708 administered by IV injection
  Interventions: Drug: LY4066708
- Part B Cohort 1: Multiple-Ascending Dose (MAD)- LY4066708 (Experimental): LY4066708 administered by IV injection
  Interventions: Drug: LY4066708
- Part B Cohort 2: MAD- LY4066708 (Experimental): LY4066708 administered by IV injection
  Interventions: Drug: LY4066708
- Part B Cohort 3: MAD- LY4066708 (Experimental): LY4066708 administered by IV injection
  Interventions: Drug: LY4066708
- Part B Cohort 4: MAD- LY4066708 (Experimental): LY4066708 administered by IV injection
  Interventions: Drug: LY4066708
- Placebo (Placebo Comparator): Placebo administered by IV injection
  Interventions: Drug: Placebo
- Placebo- Part A Cohort 3A and Part A Cohort 3B. (Placebo Comparator): Placebo administered by SC injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY4066708 — Administered IV
  Arms: Part A Cohort 1: Single-Ascending Dose (SAD)- LY4066708; Part A Cohort 2: SAD- LY4066708; Part A Cohort 4: SAD- LY4066708; Part A Cohort 5: SAD- LY4066708; Part A Cohort 5A: SAD- LY4066708; Part A Cohort 6: SAD- LY4066708; Part A Cohort 6A: SAD- LY4066708; Part B Cohort 1: Multiple-Ascending Dose (MAD)- LY4066708; Part B Cohort 2: MAD- LY4066708; Part B Cohort 3: MAD- LY4066708; Part B Cohort 4: MAD- LY4066708
Drug: Placebo — Administered IV
  Arms: Placebo
Drug: LY4066708 — Administered SC
  Arms: Part A Cohort 3A: SAD- LY4066708; Part A Cohort 3B: SAD- LY4066708
Drug: Placebo — Administered SC
  Arms: Placebo- Part A Cohort 3A and Part A Cohort 3B.

SUMMARY:
The main purpose of this study is to explore the safety and any side effects of LY4066708 in healthy participants. The study will also measure how much LY4066708 gets into the bloodstream and the central nervous system and how long it takes the body to remove it. The study will last up to 24 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Japanese Participants Only: To qualify as a participant of first-generation Japanese origin, the participant, the participant's biological parents, and all the participant's biological grandparents must be of exclusive Japanese descent and born in Japan.
* Chinese Participants Only: To qualify as Chinese for the purpose of this study, all 4 of the participants' biological grandparents must be of exclusive Chinese descent and born in China, Hong Kong, Macau, or Taiwan.
* Have a body mass index (BMI) at the time of screening within the range 18.5 to 30 kilogram per meter squared (kg/m²) (inclusive).
* Participants assigned female at birth (AFAB) not of childbearing potential and participants assigned male at birth (AMAB) willing to practice effective contraception throughout the study may participate.
* Willingness to undergo study procedures which may include repeated lumbar punctures

Exclusion Criteria:

* Are individuals of childbearing potential (IOCBP). Notwithstanding their IOCBP status, participants AFAB are excluded if they are breastfeeding.
* A history of additional risk factors for Torsades de Pointes (for example, heart failure, hypokalemia, family history of Long QT Syndrome).
* The use of concomitant medications that prolong the QT/QTc interval.
* Have known allergies to LY4066708 or any components of the formulation, or history of allergic reactions to any transferrin receptor (TfR) antibodies.
* Have participated, within the 3 months of screening, in a clinical trial involving a study intervention (other than the study intervention used in this study). If the previous investigational product has a long half-life (t½), 3 months or 5 half-lives (whichever is longer) should have passed.
* Are persons who have previously completed or withdrawn from this study and have previously received the study intervention. This exclusion criterion does not apply to subjects who are allowed to rescreen prior to randomization.
* Have a 12-lead electrocardiogram (ECG) abnormality at screening that, in the opinion of the investigator, increases the risks associated with participating in the study, or may confound ECG data analysis.
* Show evidence of hepatitis C and/or positive hepatitis C antibody.
* Current infection with hepatitis B virus (HBV) or evidence of past infection with HBV, that is, positive for Hepatitis B surface antigen (HBsAg) or Hepatitis B core total antibody (anti-HBc).
* A marked baseline prolongation of time from the start of the Q wave to the end of the T wave/ corrected QT interval (QT/QTc) interval (for example, repeated demonstration of a corrected time from the start of the Q wave to the end of the T wave interval - Fridericia formula (QTcF) interval greater than 450 ms).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Part A: Number of Participants with One or More Serious Adverse Events (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Week 12
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Adverse Events module
Part B: Number of Participants with One or More Serious Adverse Events (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Screening to Day 22
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Adverse Events module

SECONDARY OUTCOMES:
Part A: Pharmacokinetics (PK)- Area Under the Plasma Concentration Versus Time Curve (AUC0-168) | Predose up to day 15
  To evaluate PK after a single dose of LY4066708
Part B: Pharmacokinetics (PK)- AUC0-168 | Day 1 up to day 7
  To evaluate PK after multiple doses of LY4066708
Part A: Pharmacokinetics (PK)- Maximum Observed Drug Concentration (Cmax) | Predose up to day 15
  To evaluate PK after a single dose of LY4066708
Part B: Pharmacokinetics (PK)- Cmax | After dose 3, up to day 64
  To evaluate PK after a single dose of LY4066708

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Fortrea Clinical Research Unit, Holbeck, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No